CLINICAL TRIAL: NCT06277687
Title: Exploratory Study on the Application of Virtual Augmented Reality Combined With Finder in Preoperative Anterolateral Thigh Flap Perforator Positioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Song Fan, MD, Associate Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SYSKY-2024-023-02
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Blood Vessel Perforation
Keywords: anterolateral thigh flap; Finder; Virtual Augmented Reality; computerized tomography; color doppler ultrasound

STUDY DESIGN:
Intervention Model Description: After performing CTA examination, input the CTA data into Cinematic Anatomy reconstruction software to analyze blood vessels, muscles and other tissues are reconstructed in three dimensions. Before the operation, the Finder is used to restore the position of the thigh during CTA examination. The Hololens is used to match the reconstructed three-dimensional image with the Finder and the thigh. Before the operation, the pedicles of the descending branches of the lateral arteries and the perforating vessels are marked on the skin of the thigh to achieve the positioning and marking of the perforating branches.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- perforator localization (Experimental): Virtual Augmented Reality combined with Finder and Color Doppler Ultrasound were used to locate the perforating branch of the descending branch of the lateral circumflex femoral artery, and the position of the perforator was compared with real perforator respectively during the operation.
  Interventions: Diagnostic Test: Virtual Augmented Reality Combined With Finder

INTERVENTIONS:
Diagnostic Test: Virtual Augmented Reality Combined With Finder — After CT examination, the computer carried out three-dimensional reconstruction of blood vessels, and input the CTA data into Cinematic Anatomy reconstruction software to analyze blood vessels, Muscles and other tissues are reconstructed in three dimensions. Before the operation, the Finder is used to restore the position of the thigh during CTA examination. The Hololens is used to match the reconstructed three-dimensional image with the perforator locator and the thigh. Before the operation, the pedicles of the descending branches of the lateral arteries and the perforating vessels are marked on the skin of the thigh to achieve the positioning and marking of the perforating branches.
  Other Names: Color Doppler ultrasound

SUMMARY:
Oral and maxillofacial region is an important anatomical part of human body, responsible for chewing, swallowing, language, expression, breathing and other physiological functions. The tissue defects in this area not only seriously affect the physiological function, but also lead to facial deformity and aesthetic damage, affecting the quality of life of patients. The anterolateral thigh flap has become one of the main methods for defect repair due to its large tissue volume and high survival rate, and one of the key steps to ensure a high survival rate is the location of the perforator. How to find the perforator more accurately by improving the detection scheme or locating the perforator according to the anatomical structure, and guide the preparation and cutting of the flap, is the main direction of current research. This study intends to conduct a exploratory study on perforator localization of flap , and explore its effectiveness and accuracy through sensitivity and specificity.

In this study, a total of 24 patients with maxillofacial defects caused by tumors, trauma and other reasons requiring anterolateral femoral flap repair were included, and the perforator branch of femoral anterolateral flap was positioned preoperatively by Virtual augmented reality combined with perforator positioning device and color Doppler ultrasound. After the anterolateral thigh flap was prepared, the incision was closed in the donor area of the leg, and the flap was transplanted free to the maxillofacial defect area for repair. The sensitivity, specificity, positive predictive value, negative predictive value, distance difference and odds ratio of the two methods were calculated respectively, and the differences of each evaluation index between the two groups were compared, mainly to evaluate the sensitivity and specificity between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with oral and maxillofacial defects caused by malignant tumors or trauma require anterior lateral femoral skin flap repair after surgery
2. There is no history of leg trauma and surgery is feasible
3. No clinically significant positive signs were found in physical examination
4. No chronic or current illnesses such as heart, liver, pancreas, spleen, kidney, digestive tract, respiratory, blood, nervous system, etc
5. No abnormalities found in electrocardiogram (ECG) and X-ray film
6. Hepatitis B surface antigen (HBSAg), anti hepatitis C antibody (anti HCV), anti human immunodeficiency virus antibody (anti HIV), and negative Treponema pallidum (TP)
7. No clinically significant abnormalities were found in vital signs, blood routine, urine routine, blood biochemistry, and blood pregnancy tests
8. The patient voluntarily participated in this study and signed an informed consent form

Exclusion Criteria:

1. Have a history of leg injury or surgery
2. Significant abnormalities in blood routine, heart, lung, liver, and kidney functions, insufficient compensatory function, or severe systemic diseases
3. Pregnant or lactating women, or those planning to conceive within six months
4. Individuals with a history of mental illness who cannot cooperate with the examination
5. Individuals with allergic constitution or known allergies to contrast agent ingredients
6. The patient or guardian refuses to sign a written consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity | during the operation
  The percentage of actual perforating branches that are correctly determined as the perforating branches according to this research method (true positive rate) is calculated as follows: number of true positive perforations /(number of true positive perforations + number of false negative perforations) =TP/(TP+FN)
Specificity | during the operation
  The percentage of actual no perforations correctly judged as no perforations according to this research method (true negative rate) is calculated as follows: true negative number /(true negative perforations + false positive perforations) =TN/(TN+FP)

SECONDARY OUTCOMES:
positive predictive value | during the operation
  The proportion of true positivity in the number of positive perforations determined by this research method reflects the probability that the subject does have perforations when the diagnostic method to be evaluated is determined to be positive. The calculation formula is as follows: PV+ = number of true positive perforations/total number of perforations =TP/(TP+FP)
negative predictive value | during the operation
  The proportion of true negative in the number of negative non-penetrating counts determined by the research method; If the diagnostic method to be evaluated is judged negative, the probability that the subject has no negative is calculated as follows: PV- = number of true negative penetrations/total number of controls =TN/(FN+TN)
Youden Index | during the operation
  Defined as the total ability to find the correct perforating branches and to judge the absence of perforating branches, is the sum of sensitivity and specificity minus 1

CONTACTS AND LOCATIONS:
Overall Officials: Song Fan, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guanzhou, Guangdong, China